CLINICAL TRIAL: NCT00335179
Title: Double-Blind, Vehicle-Controlled Study to Evaluate Cellular and Molecular Events During Four Weeks of Treatment for Actinic Keratosis With Aldara (Imiquimod) Cream, 5%
Brief Title: Cellular and Molecular Events During Treatment of Actinic Keratosis With Imiquimod 5% Cream
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Graceway Pharmaceuticals, LLC (Industry)
Responsible Party: James Lee, MD, Graceway Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1467-IMIQ
Record Dates: First submitted 2006-06-08; First posted 2006-06-09 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Actinic Keratosis
Keywords: Actinic keratosis; AK; imiquimod; confocal microscopy; gene microarray
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imiquimod cream (Active Comparator): Imiquimod 5% cream containing 12.5 mg of imiquimod per 250 mg of cream Applied 3 times per week for 4 weeks
  Interventions: Drug: Aldara (imiquimod 5% cream)
- Vehicle cream (Placebo Comparator): Vehicle cream 250 mg Applied 3 times per week for 4 weeks
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: Aldara (imiquimod 5% cream) — Imiquimod 5% cream containing 12.5 mg of imiquimod per 250 mg of cream
  Other Names: imiquimod cream
  Arms: Imiquimod cream
Drug: Vehicle cream — Vehicle cream in 250 mg
  Other Names: placebo cream
  Arms: Vehicle cream

SUMMARY:
Treatment of actinic keratosis with imiquimod cream is expected to cause changes in the genes that are turned on, and turned off, by skin cells. Some of the drug induced changes in skin cells should also be visible using a special microscope. This study examines both types of changes.

DETAILED DESCRIPTION:
The primary objective of this study was to assess apoptosis by examining the gene expression profiles of actinic keratosis (AK) lesions that were treated with imiquimod 5% cream or vehicle cream once daily 3 times per week for 4 weeks. Secondary objectives were to assess the utility of confocal microscopy (CM) to visually track cellular response to treatment with study cream compared with clinical and histological evaluations, and to evaluate the safety of treatment with imiquimod in subjects with AK on the balding scalp.

ELIGIBILITY:
Inclusion Criteria:

* Have actinic keratoses on balding scalp
* Discontinuation of tanning bed use
* Discontinuation of moisturizers
* Avoidance of retinol products

Exclusion Criteria:

* Uncontrolled, clinically significant medical condition
* Dermatologic disease other than actinic keratosis in treatment area

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2003-01; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Gene expression profiling of treated lesions | weeks 1, 2, and 4, and at 4 weeks post-treatment

SECONDARY OUTCOMES:
Confocal microscopic evaluation before, during and post treatment | weeks 1, 2, 4 and at 4 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: TC Meng, MD, Study Director — Graceway Pharmaceuticals
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

REFERENCES:
- [Background] Torres A, Storey L, Anders M, Miller RL, Bulbulian BJ, Jin J, Raghavan S, Lee J, Slade HB, Birmachu W. Microarray analysis of aberrant gene expression in actinic keratosis: effect of the Toll-like receptor-7 agonist imiquimod. Br J Dermatol. 2007 Dec;157(6):1132-47. doi: 10.1111/j.1365-2133.2007.08218.x. Epub 2007 Oct 18. PMID 17944981
- [Background] Torres A, Storey L, Anders M, Miller RL, Bulbulian BJ, Jin J, Raghavan S, Lee J, Slade HB, Birmachu W. Immune-mediated changes in actinic keratosis following topical treatment with imiquimod 5% cream. J Transl Med. 2007 Jan 26;5:7. doi: 10.1186/1479-5876-5-7. PMID 17257431